CLINICAL TRIAL: NCT03486795
Title: Effect of Dual Site-Dual Channel Non-invasive Brain Stimulation for Recovery of Motor Function in Healthy Subjects
Brief Title: Dual Site-Dual Channel Non-invasive Brain Stimulation for Motor Function in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-08-124-C
Record Dates: First submitted 2018-03-22; First posted 2018-04-03 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2018-03

CONDITIONS: Healthy
Keywords: transcranial direct current stimulation; motor function

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dual stimulation (Experimental): 1. anodal stimulation on right primary motor cortex and cathodal stimulation on left primary motor cortex
  2. anodal stimulation on right premotor cortex and cathodal stimulation on left supraorbital area
  Interventions: Device: M1 stimulation
- M1 stimulation (Experimental): anodal stimulation on right primary motor cortex and cathodal stimulation on left primary motor cortex
  Interventions: Device: M1 stimulation
- PMC stimulation (Experimental): anodal stimulation on right premotor cortex and cathodal stimulation on left supraorbital area
  Interventions: Device: PMC stimulation
- Sham stimulation (Sham Comparator): Sham stimulation
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: M1 stimulation — stimulating primary motor cortex with anodal stimulation on right primary motor cortex and cathodal stimulation on left primary motor cortex
  Arms: Dual stimulation; M1 stimulation
Device: PMC stimulation — stimulating premotor cortex with anodal stimulation on right premotor cortex and cathodal stimulation on left supraorbital area
  Arms: PMC stimulation
Device: Sham stimulation — sham stimulation over both primary motor cortex and premotor cortex
  Arms: Sham stimulation

SUMMARY:
The aim of this study is to investigate the effect of dual site-dual channel non-invasive brain stimulation for recovery of motor function in healthy subjects. Simultaneous dual site-dual channel stimulation was applied by using two sets of transcranial direct current stimulation devices. All subjects will go through four conditions of transcranial direct current stimulation with for 30 minutes. Four conditions are 1) Dual stimulation: i) anodal stimulation on right primary motor cortex and cathodal stimulation on left primary motor cortex, ii) anodal stimulation on right premotor cortex and cathodal stimulation on left supraorbital area. 2) M1 stimulation: anodal stimulation on right primary motor cortex and cathodal stimulation on left primary motor cortex; 3) PMC stimulation: anodal stimulation on right premotor cortex and cathodal stimulation on left supraorbital area. 4) sham stimulation

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects with age over 19 years old

Exclusion Criteria:

* history of disorders involving central nervous system
* patients with severe medial or psychiatric disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Changes in motor evoked potential | Baseline and after intervention (approximately 30 minutes)
  measure the motor threshold and amplitude of motor evoked potential in first dorsal interosseous muscle

SECONDARY OUTCOMES:
Changes in sequential motor task | Baseline and after intervention (approximately 30 minutes)
  measures motor functional and dexterity of hand

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided